CLINICAL TRIAL: NCT03129854
Title: A Randomized Study of Androgen Deprivation Therapy Versus Androgen Deprivation Therapy Plus Prostate Cryotherapy in the Treatment of Patients With Primary Diagnosed Metastatic Prostate Cancer
Brief Title: Androgen Deprivation Therapy (ADT) Versus ADT Plus Prostate Cryotherapy for Metastatic Prostate Cancer (mPCa)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yonghong Li, Principal Investigator, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YoLi
Record Dates: First submitted 2017-04-16; First posted 2017-04-26 (Actual); Last update posted 2019-06-07 (Actual); Status verified 2019-06

CONDITIONS: Prostate Cancer Metastatic
Keywords: prostate cancer; metastatic; cryotherapy; ADT
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Intervention Model Description: One group receive standard of care ADT continually. Another group receive ADT plus prostate cryotherapy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Prostate cryotherapy plus ADT
  Interventions: Device: prostate cryotherapy
- control group (No Intervention): standard of care ADT continually

INTERVENTIONS:
Device: prostate cryotherapy — prostate cryotherapy added to experimental group within 6 months of ADT
  Other Names: prostate cryoablation
  Arms: experimental group

SUMMARY:
Patients with primary diagnosed metastatic prostate cancer are randomly divided into two groups. One group receive standard of care ADT continually. Another group receive ADT plus prostate cryotherapy. Patients are followed up until their death or withdraw from this study due to other reasons. The primary endpoint of this study is prostate cancer Progression-Free Survival. The secondary endpoint is overall survival, prostate cancer specific survival and health-related quality of life.

DETAILED DESCRIPTION:
Ages Eligible for Study: 18 Years and older.

Genders Eligible for Study: Male.

Accepts Healthy Volunteers: No.

ELIGIBILITY:
Inclusion Criteria:

* Have histologically diagnosed prostate cancer
* Metastatic disease diagnosed by CT scan, MRI scan or bone scan. M stage M1a or M1b according to 2010 American joint Committee on Cancer (AJCC) stage system
* Be willing and able to provide written informed consent/assent for the trial
* Eastern Cooperative Oncology Group (ECOG) performance scale status of 0 or 1
* Calculator of overall mortality risk at 3 years less than 70%( Eur Urol. 2016 May 9. pii: S0302-2838(16)30141-5. )
* Time interval between hormonal therapy and randomization less than 6 months
* Can tolerate general anesthesia and cryosurgery
* Demonstrate adequate organ function

Exclusion Criteria:

* According to the doctor's judgment, the patients had any serious illness or other clinical conditions, can't safely undergo the clinical research, any other serious diseases or clinical situation is not limited to the items listed below:

  * Infection ≥ grade 2 according to National Cancer Institute on the common terminology criteria for adverse events (NCI-CTCAE) version 4.03,
  * Heart failure (New York heart group NYHA) III or IV,
  * Crohn's disease or ulcerative colitis,
  * Fecal incontinence,
  * Substance abuse, medical, psychological or social problems that may interfere with the evaluation of the results of this study,
  * The presence of any unstable disease or clinical condition, potential harm to the safety of the subject or influence the subject's compliance.
* Other malignancies (within 5 years), except for non melanoma skin cancer. Patients with other malignancies who survived with effective treatment and randomized to have no evidence of cancer for more than 5 years were allowed to participate in the study
* Treatment of prostate cancer other than hormonal therapy (except bisphosphonate therapy for bone metastases)
* After 6 months of hormonal treatment, the prostate volume greater than 55ml

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Gender identity
Enrollment: 250 (Estimated)
Dates: Start 2017-03-29 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Prostate Cancer Progression-Free Survival | through study completion, an average of 48 months
  Prostate Cancer Progression-Free Survival (PFS), from beginning of ADT to progression of prostate cancer

SECONDARY OUTCOMES:
Overall Survival | through study completion, an average of 60 months
  Overall Survival (OS), from beginning of ADT to death
prostate cancer specific survival | through study completion, an average of 60 months
  prostate cancer specific survival (CSS), from beginning of ADT to death from prostate cancer
Functional Assessment of Cancer Therapy-Prostate | through study completion, an average of 48 months
  Functional Assessment of Cancer Therapy-Prostate (FACT-P), From beginning of ADT to death

CONTACTS AND LOCATIONS:
Overall Officials: Minghuang Hong, MD, Study Director — Sun Yat-sen University
Locations (1):
- Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Loppenberg B, Dalela D, Karabon P, Sood A, Sammon JD, Meyer CP, Sun M, Noldus J, Peabody JO, Trinh QD, Menon M, Abdollah F. The Impact of Local Treatment on Overall Survival in Patients with Metastatic Prostate Cancer on Diagnosis: A National Cancer Data Base Analysis. Eur Urol. 2017 Jul;72(1):14-19. doi: 10.1016/j.eururo.2016.04.031. Epub 2016 May 9. PMID 27174537
- [Background] Culp SH, Schellhammer PF, Williams MB. Might men diagnosed with metastatic prostate cancer benefit from definitive treatment of the primary tumor? A SEER-based study. Eur Urol. 2014 Jun;65(6):1058-66. doi: 10.1016/j.eururo.2013.11.012. Epub 2013 Nov 20. PMID 24290503
- [Background] Babaian RJ, Donnelly B, Bahn D, Baust JG, Dineen M, Ellis D, Katz A, Pisters L, Rukstalis D, Shinohara K, Thrasher JB. Best practice statement on cryosurgery for the treatment of localized prostate cancer. J Urol. 2008 Nov;180(5):1993-2004. doi: 10.1016/j.juro.2008.07.108. Epub 2008 Sep 25. No abstract available. PMID 18817934